CLINICAL TRIAL: NCT00290108
Title: The Influence of Injection Rate on EEG Propofol Peak Effect as Measured by Bispectral Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 257/99
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2006-02-10 (Estimated); Status verified 1998-06

CONDITIONS: Elective Surgery; Healthy
Keywords: BIS; Propofol; hemodynamic; pharmacokinetic
MeSH Terms: interventions — Propofol

INTERVENTIONS:
Drug: Propofol

SUMMARY:
The aim of the present study was to investigate whether injection rate of propofol has an influence on its maximum effect.

DETAILED DESCRIPTION:
The clinical daily routine indicates that slowing the rate of administration of propofol can lead to a reduction of up to 50% in the dose of propofol required to achieve the onset of a clinical endpoint of anesthesia (i.e. loss of consciousness) when titrating to effect. Therefore, it has been concluded that a slow injection requires a smaller dose of propofol as the graded effect is weakened by fast injection. This conclusion contradicts pharmacologic considerations, that a fast injection would lead to a higher peak concentration and in consequence, to a higher peak effect at the effect side, the brain.

The present study was designed to measure the Electroencephalogram (EEG) peak effect of a propofol bolus (2 mg/kg) injected with different infusion rates.

Although it is known that propofol has cardiovascular effects, the influence of injection rate on these cardiovascular changes is less clear. Others found that faster injection rates of propofol caused greater reductions in blood pressure. Other similar studies have shown no difference in blood pressure for different injection rates. An additional aim of this study was therefore to investigate the influence of different injection rates on hemodynamic parameters.

ELIGIBILITY:
Inclusion criteria:

* American Society of Anesthesiologists (ASA) physical status 1-3
* scheduled for elective surgery under general anesthesia.

Exclusion criteria:

* emergency surgery
* obesity
* indication for rapid sequence induction
* drugs that affect the central nervous system
* history of alcohol or drug abuse
* neurological or psychiatric diseases
* contraindications against the use of propofol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99
Dates: Start 2003-03; Study Completion 2003-12

PRIMARY OUTCOMES:
maximum hypnotic effect as indicated by the minimum BIS value.

SECONDARY OUTCOMES:
time to loss of consciousness
time to loss of eye lash reflex
time to BISmin
BIS at LOC
BIS at LOL
BIS 30 seconds after LOC

CONTACTS AND LOCATIONS:
Overall Officials: Eberhard Kochs, MD, Study Chair
Locations (1):
- Technische Universität München, Klinikum rechts der Isar, Department of Anesthesiology, Munich, Bavaria, Germany